CLINICAL TRIAL: NCT06877325
Title: Synergistic Effects of Traditional Chinese Medicine Practices and Pelvic Floor Muscle Training on Postpartum Stress Urinary Incontinence
Brief Title: Synergistic Effects of Traditional Chinese Medicine Practices and Pelvic Floor Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangxi College for Preschool Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCPI2022
Record Dates: First submitted 2025-02-27; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Maternal Stress
MeSH Terms: interventions — Qigong

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pelvic floor muscle training (Experimental)
  Interventions: Behavioral: PFMT
- Qigong with pelvic floor muscle training (Experimental)
  Interventions: Behavioral: QGPFMT
- Qigong (Experimental)
  Interventions: Behavioral: Qigong

INTERVENTIONS:
Behavioral: PFMT — The training is divided into three phases. The first phase is the foundation phase (Weeks 1-4), which primarily activates the pelvic floor muscles. Strengthening Phase (Weeks 5-8): Builds muscular endurance and control by increasing contraction duration. Consolidation Phase (Weeks 9-12): Enhances overall stability and strength through functional movements.
  Arms: Pelvic floor muscle training
Behavioral: QGPFMT — The training is divided into three phases: Foundation Phase (Weeks 1-4): Focuses on breath regulation and activation to promote energy flow and awaken the pelvic floor muscles. Strengthening Phase (Weeks 5-8): Combines core stability training to enhance muscle strength and flexibility. Consolidation Phase (Weeks 9-12): This phase strengthens core control while incorporating standing meditation and breathing exercises to harmonize body and mind, improving overall stability and endurance.
  Arms: Qigong with pelvic floor muscle training
Behavioral: Qigong — The training is divided into three phases. The first phase (Weeks 1-4) focuses on breathing regulation and relaxation to enhance blood circulation and promote body recovery. Strengthening Phase (Weeks 5-8): Utilizes "Dao Yin" techniques to improve flexibility and stimulate energy flow. Consolidation Phase (Weeks 9-12): Emphasizes overall enhancement and core strengthening and incorporates extended deep breathing meditation to harmonize body and mind.
  Arms: Qigong

SUMMARY:
This study was conducted within a randomized controlled trial framework using a double-blind design. Participants were assigned to one of three intervention groups: the Pelvic Floor Muscle Training group (PFMT), the Pelvic Floor Muscle Training combined with the Qigong group (PFMTQG), and the Qigong Practice group (QG). Randomization was performed using a random number table. Professional trainers implemented the intervention programs. Researchers conducted a 12-week intervention study, with training sessions held thrice weekly. During the trial, participants agreed not to engage in other forms of physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-35 years.
* Within 12 months postpartum.
* Diagnosed with mild to moderate SUI.
* Physically capable of participating in mild to moderate exercise.
* Provided written informed consent.

Exclusion Criteria:

* Severe pelvic floor dysfunction.
* Systemic health conditions that contraindicate physical activity.
* Pregnant at the time of recruitment or planning pregnancy during the study
* Prior structured training in Qigong or PFMT.
* Ongoing physiotherapy for pelvic floor health.
* Participation in other urinary incontinence research.
* Inability to provide informed consent due to cognitive or language barriers.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Incontinence Episode Frequency | Month 3
  Incontinence Episode Frequency (IEF) will be measured using a 72-hour bladder diary maintained by participants. Participants will be provided with a structured bladder diary template, which includes columns for recording each instance of urine leakage, the associated activity (e.g., coughing, sneezing, physical exertion), and the approximate volume of leakage (if subjectively estimable). The frequency of urine leakage episodes will be calculated by averaging the total number of incidents recorded over the three days at each assessment point. The 72-hour urinary incontinence episode values will represent the total number of leakage incidents observed across the three days and will be used to evaluate changes in IEF over time.
1-hour Pad Test | Month 3
  Urine leakage will be objectively quantified using the 1-hour pad test, conducted at the same time points as the bladder diary assessments. Participants will be provided with pre-weighed absorbent pads and instructed to wear them for a continuous 1-hour period. During this time, participants will be asked to drink 500 ml of plain water over 15 minutes and perform normal activities, including simple walking for the next 30 minutes. In the last 15 minutes, participants will be instructed to perform the standard ICS provocation exercises in a private area. If a participant is found to have vaginal bleeding or excessive vaginal discharge, the test will be postponed and rescheduled for a later date. After the 1-hour period, participants will seal the pads in provided plastic bags and return them to the study site. Trained assessors will measure the weight difference between the pre- and post-use pads using a precision digital scale .

SECONDARY OUTCOMES:
Pelvic Floor Muscle Assessment | Month 3
  Pelvic floor muscle function will be assessed using a Peritron 9300V perineometer (Cardio Design Pty Ltd., Melbourne, Australia), a device widely used in clinical and research settings for measuring intravaginal pressure. To standardize measurements, participants will be asked to empty their bladder prior to the test, and the procedure will be thoroughly explained by the assessor to ensure understanding and comfort. Participants will undergo the assessment in a semi-recumbent position with knees bent and feet flat on the examination table. A sterile, single-use intravaginal pressure sensor will be lubricated with a water-based gel and inserted to ensure proper placement and participant comfort. During the assessment, participants will perform three maximal voluntary pelvic floor muscle contractions, each held for 5 seconds, with 10-second rest intervals between contractions to avoid fatigue. The highest pressure recorded from the three attempts will be used for analysis.
Incontinence Impact Questionnaire-7 | Month 3
  This tool is specifically designed to evaluate the effects of urinary incontinence on participants' daily lives, encompassing physical, emotional, and social domains. The IIQ-7 is a subset of the full Incontinence Impact Questionnaire, developed to measure the impact of urinary incontinence on women's quality of life in a concise format. It consists of seven items addressing the extent to which urinary leakage interferes with: physical activities, social interactions and emotional well-being. The total score ranges from 0 to 28, with higher scores indicating a greater negative impact on quality of life.
Urinary Distress Inventory-6 | Month 3
  The UDI-6 is a short-form version of the Urinary Distress Inventory and evaluates symptom-related distress associated with urinary incontinence. The six items target: urinary urgency, frequency, urinary leakage and bladder control issues.
  Each item is scored on a 4-point Likert scale ranging from 0 = Not at all to 3 = Greatly. Total scores range from 0 to 24, with higher scores reflecting greater symptom distress.
Psychological Well-being Assessment | Month 3
  Psychological well-being will be evaluated using the Perceived Stress Scale (PSS), a validated and widely used questionnaire designed to assess perceived stress levels over the past month. The PSS consists of 10 items, each reflecting an aspect of stress perception, such as feelings of unpredictability, uncontrollability, and being overwhelmed. Participants will rate their responses on a 5-point Likert scale, where 0 = never and 4 = very often, based on their experiences in the preceding month. Total scores range from 0 to 40, with higher scores indicating greater levels of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No